CLINICAL TRIAL: NCT04290910
Title: A Pilot Study Evaluating the Clinically Managed Weight Loss Program At the Wellness Institute At Seven Oaks General Hospital
Brief Title: A Pilot Study Evaluating a Clinically Managed Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS22267 (H2018:401)
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: pilot study; program evaluation; nutrition; exercise; psychology
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Weight Loss Program (Experimental): Single arm, all participants receive the weight loss program
  Interventions: Behavioral: Weight Loss Program

INTERVENTIONS:
Behavioral: Weight Loss Program — There are three components of the intervention, this includes: psychology, nutrition, and physical activity. For the psychological portion, a therapist will assess the participant at baseline to determine if there are barriers associated with making lifestyle changes. For nutrition, the dietitian will assess the participant and create a meal plan based on their nutritional needs and guide the participant to reaching their nutritional goals. The psychological and nutrition portion may be interchangeable depending on the participants needs. For physical activity, the personal trainer will assess the participant and create an exercise plan that consists of resistance training and weight bearing exercises suitable for the participant while also guiding the participant to reach their exercise goals.

SUMMARY:
This is a pilot study evaluating a clinically managed weight loss program. The program consists of a 17-week weight loss program which involves a multidisciplinary team where personalized interventions are given to participants from the team based on the participants goals.

DETAILED DESCRIPTION:
The clinically managed weight loss program is managed by a clinical team including a Program Manager, Registered Dietitians, Canadian Society of Exercise Physiology-Certified Personal Trainers, Clinical Psychology Associate or Cognitive Behavioural Therapist, and a Physician. The team will collaborate together to prescribe a plan best suited for the participants' needs with the focus on lifestyle changes, such as, sleep, mental health, and behaviours. Outcome measures will be collected as part of the pilot study, such as, anthropometric measurements and body composition, cardiovascular assessment, clinical chemistry, physical activity, nutrition, and behaviour and health screening questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or female, aged 18 years or above.
* Are overweight or obese (BMI over 24.9)

Exclusion Criteria:

- Female participant who is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Body Weight Loss | 4 months
  Weight will be measured in kg to the nearest 0.1 kg using a InBody 570 scale

SECONDARY OUTCOMES:
Changes in Quality of Life | 4 months
  Quality of life will be measured through the SF-36 quality of life questionnaire. The SF-36 measures nine areas: physical functioning, role functioning (emotional), role functioning (physical), energy/fatigue, emotional well-being, social functioning, pain, general health, and health change. A higher score indicate greater levels of quality of life.
Changes in Sleep Quality | 4 months
  Sleep will be measured through the Pittsburgh Sleep Quality Index questionnaire. The Pittsburgh Sleep Quality Index questionnaire measures the quality and pattern of sleep in adults, and includes seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. A score of 5 or less is indicated as good sleep quality where a score of 6 or more is indicated as poor sleep quality.

OTHER OUTCOMES:
Attendance | 4 months
  Attendance will be measured by checking if participants have attended each appointment with the health care professional as implemented by the program.
Intervention Adherence | 4 months
  Intervention adherence will be measured by checking if participants have attended each appointment with the health care professional as implemented by the program. If the participant has attended 80% or more of their appointments, this would be classified as good intervention adherence to the program.
Waist Circumference | 4 months
  Waist circumference in cm will be measured in triplicate, to the nearest 0.1 cm at the umbilicus, between the last rib and iliac crest using a fibreglass tape measured by an exercise professional.
Body fat percentage | 4 months
  The InBody 570 Body Composition Analyzer will measure body fat percentage by bioelectrical impedance.
Lean mass percentage | 4 months
  The InBody 570 Body Composition Analyzer will measure lean mass percentage by bioelectrical impedance.
Systolic Blood Pressure | 4 months
  Systolic blood pressure in mmHg is measured in triplicate, on the non-dominant arm in a sitting position by an exercise professional using a validated oscillometric blood pressure monitor.
Diastolic Blood Pressure | 4 months
  Diastolic blood pressure in mmHg is measured in triplicate, on the non-dominant arm in a sitting position by an exercise professional using a validated oscillometric blood pressure monitor.
Heart Rate | 4 months
  Heart rate in beats per minute is measured in triplicate, on the non-dominant arm in a sitting position by an exercise professional using a validated oscillometric blood pressure monitor.
Total cholesterol | 4 months
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol concentration in mmol/L according to their established protocols.
High density lipoprotein cholesterol | 4 months
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the high density lipoprotein cholesterol concentration in mmol/L according to their established protocols.
Low density lipoprotein cholesterol | 4 months
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the low density lipoprotein cholesterol concentration in mmol/L according to their established protocols.
Triglyceride | 4 months
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the triglyceride concentration in mmol/L according to their established protocols.
total cholesterol and high density lipoprotein cholesterol ratio | 4 months
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the total cholesterol and high density lipoprotein cholesterol ratio according to their established protocols.
Hemoglobin A1C | 4 months
  Diagnostic Services of Manitoba will collect and process the participants blood samples and measure the hemoglobin A1C as a percentage according to their established protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Wellness Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No